CLINICAL TRIAL: NCT02390271
Title: Cardiac Coherence Training to Reduce Anxiety in Remitted Schizophrenia
Brief Title: How Reducing Anxiety in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: m trousselard
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- emotion focused therapy training CCT (Experimental): The general training includes in an individual adjusted way the following techniques: biofeedback-assisted breathing classes that erase negative emotion involving the cardiac and limbic neural pathways, control one's own and other's emotions, mastering positive cognition and enhance self-concept, anchoring positive memories, learning how to recognize psychological reversal in others
  Interventions: Other: emotion focused therapy training

INTERVENTIONS:
Other: emotion focused therapy training — The Cardiac Coherence Training (CCT) incorporates a series of emotion-refocusing and restructuring techniques involving the use of biofeedback to control heart rate variability
  Other Names: Cardiac Coherence Training

SUMMARY:
Introduction: Health care that addresses the emotional regulation capacity of patients with schizophrenia confronted with daily stress may contribute to a less anxious life. A psycho-physiological training (cardiac coherence training; CCT) focusing on emotion regulation is known to decrease anxiety for non-clinical individuals.

Methods: the investigators performed a pilot cross sectional survey to explore the benefits of CCT for clinically stable patients with schizophrenia. Ten patients were enrolled in the program consisting in height to twelve weekly one hour session program during a 2-month follow-up. Standardised questionnaires were used before and after the intervention assessing anxiety, well-being outcomes, and how patients deal with stress and stressors.

DETAILED DESCRIPTION:
Ten subjects, five women and five men, all volunteers, were included in the study. The patients were all clients of the rehabilitation center for psychotic disorders (Le Vinatier hospital) situated in Lyon, France. Criteria for entry into the study included: a Diagnostic and Statistical Manual of Mental Disorder-4 diagnosis of schizophrenia as confirmed by the Mini International Neuropsychiatric Interview for DSM-IV (MINI); age between 18 and 65; being clinically stable (i.e. not having required hospitalization or increases in medication as a result of an exacerbation of acute symptoms over the previous three months.

All subjects completed a set of "paper and pencil" standardized assessments at pre-intervention and immediately after the end of the intervention.

Trait and State anxiety was assessed using the French version of the Spielberger State-Trait-Anxiety Inventory (S-STAI).

Three questionnaires were used in order to evaluate the outcomes quality of life of patients. 1/ The Positive And Negative Syndrome Scale (PANSS); 2/ Patient's body/mind perceptions were assessed using mindfulness concept (Freiburg Mindfulness Inventory, FMI), and 3/ Patients' quality of life was evaluated using the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS).

One questionnaire was used to assess how patients deal with stress and stressors (the Derogatis Stress Profile, DSP).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of remitted schizophrenia

Exclusion Criteria:

* exacerbation of schizophrenic symptoms over the previous three months (hospitalization or increases in medication)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
psychometric outcome: Spielberger State Anxiety Inventory (S-STAI) | up to two months
  outcomes assessed before and after the 3-month Cardiac Coherence Training

SECONDARY OUTCOMES:
psychometric outcome: Freiburg Mindfulness Inventory (FMI) | up to two months
  outcomes assessed before and after the 3-month Cardiac Coherence Training